CLINICAL TRIAL: NCT07040813
Title: A Randomized Placebo-controlled Double-blind Phase III Trial to Investigate the Reduction of Monthly Migraine Days (MMDs) Over 12 Weeks of Treatment With CGRP mAbs and Onabotulinumtoxin A Intramuscularly Compared With CGRP mAbs and Placebo in Chronic Migraine
Brief Title: The Nordic Chronic Migraine Trial of CGRP Monoclonal Antibody and Onabotulinumtoxin A Dual Therapy Compared to CGRP mAbs Monotherapy
Acronym: NorMig
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); Sykehuset Telemark (Other Government); Sykehuset Innlandet HF (Other); Sorlandet Hospital HF (Other Government); Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT number 2024-517981-40-00
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Migraine; Chronic Migraine Headache
Keywords: Migraine; CGRP; Onabotulinumtoxin A; CGRP monoclonal antibody; Combination of CGRP mAbs and onabotulinumtoxin A
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: A randomized placebo-controlled double-blind phase III two-arm study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded study personnel will prepare the BTA/placebo with NaCl that will be administered to the participants by blinded study personnel. BTA/placebo with NaCl will be administered at 31 predeﬁned injection sites (5 units per injection; 155 units in total), in accordance with a modified version of the protocol from the Phase III REsearch Evaluating Migraine Prophylaxis Therapy 1, PREEMPT.
  To secure the blinding in the study, the four injections in the forehead will be placed in the upper frontal region whereas the injections in corrugator and procerus are kept.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGRP and placebo (Placebo Comparator): Combination of CGRP mAbs and placebo (NaCl 0.9% Braun, 0.1 ml at the same sites) in male and female participants with chronic migraine aged 18 to 70 years.
  Interventions: Drug: CGRP mAbs and placebo
- CGRP and onabotulinumtoxin A (Active Comparator): Onabotulinumtoxin A given totally 155 units at 31 sites according to modified PREEMPT or placebo (NaCl 0.9% Braun, 0.1 ml at the same sites). The treatment period is 12 weeks long.
  Interventions: Drug: CGRP mAbs and onabotulinumtoxin A

INTERVENTIONS:
Drug: CGRP mAbs and onabotulinumtoxin A — CGRP mAbs given subcutanously every 4th week and onabotulinumtoxin A 155 given once intramuscularly according to adjusted PREEMPT protocol in the 12 week period of study intervention.
  Arms: CGRP and onabotulinumtoxin A
Drug: CGRP mAbs and placebo — CGRP mAbs given subcutanously every 4th week and placebo once intramuscularly according to adjusted PREEMPT protocol in the 12 week period of study
  Arms: CGRP and placebo

SUMMARY:
Migraine is characterized by attacks of throbbing, moderate or severe headache, often associated with nausea, vomiting, and/or sensitivity to light and/or sound.

Chronic migraine, which occurs in 1-2 % of the population is characterized by 15 or more headache days/month for more than 3 months and at least 8 days/month with features of migraine headache.

The study will evaluate the efficacy of onabotulinumtoxin A when added to CGRP monoclonal antibody therapy in chronic migraine prevention. Adverse events and change in disease activity will be monitored.

Onabotulinumtoxin A and CGRP monoclonal antibody therapy are investigational drugs developed to prevent chronic migraine. Approximately 450 patients will be included from sites in Norway.

All participants will receive CGRP monoclonal antibody therapy. Additionally, the participants will be randomized to receive onabotulinumtoxin A or placebo injections.

Total study duration is 20 weeks including 3 on site visits and 3 telephone visits. After an inclusion visit the participants are registering data in an electronic headache diary using the application Brain Twin for a minimum of 4 weeks before the come to the randomization visit and the study medications are started. The duration of treatment is 12 weeks.

DETAILED DESCRIPTION:
Despite an improved understanding of migraine pathophysiology and treatment in recent years, many responders for both BTA and CGRP mAbs still experience high burden of disease. Thus, there is still a great need for further improving migraine prevention therapy. At present, there are few effective treatment alternatives for chronic migraine patients and a combination therapy of CGRP mAbs and BTA is an excellent candidate that has not previously been tested in any trial to date. The combined inhibition of CGRP release in C fibres by BTA and the receptor function blockade by CGRP mAbs directed towards the ligand or the receptor in Aδ fibres is proposed to have a synergistic effect. Several observational studies, including pooled analysis of real-world evidence, supports a combination of CGRP mAbs and BTA, but the efficacy remains to be demonstrated in randomized controlled trials. Additionally, while the cost-effectiveness of pharmacological treatments of chronic migraine in the adult population-using CGRP mAbs and BTA-have been demonstrated, the cost-effectiveness of the combination therapy needs to be clarified. As both fatigue and cognitive symptoms are important for the migraine related disability and migraine related quality of life, we will also include these aspects in the endpoint evaluations

. Hypothesis : Combination of CGRP mAbs and BTA reduces Monthly Headache Days (MHDs) in chronic migraine compared to single therapy.

In this trial of chronic migraine the efficacy of dual therapy with CGRP monoclonal antibody and onabotulinumtoxin A compared with CGRP monoclonal antibody single therapy in participants aged 18 to 70 years with chronic migraine will be studied. The primary endpoint is the reduction of Monthly Migraine Days (MMDs) over 12 weeks.

Total study duration is 20 weeks including 3 on site visits and 3 telephone visits. After an inclusion visit the participants are registering data in an electronic headache diary using the application Brain Twin for a minimum of 4 weeks before the come to the randomization visit and the study medications are started. The duration of treatment is 12 weeks.

Participants will be divided into two equal groups using electronic randomization. One group will receive one treatment with botulinum toxin A, while the other group will receive injections of placebo (saline). Unblinded study personnel will prepare botulinum toxin A/placebo which will then be administered to the participants by blinded study personnel. Onabotulinum toxin A/placebo will be administered at 31 pre-defined injection sites (0.1 ml with 5 units per injection; total 3.1 ml and 155 units), in accordance with a modified version of the Phase III REsearch Evaluating (PREEMPT) protocol. At the same time, both groups will start monthly injections of CGRP inhibitors as background medication. The choice of type of CGRP inhibitor is made by the study physician or based on national guidelines.

Participants will keep daily headache diaries throughout the study period to record headache frequency, intensity, use of reliever medication and type of headache.

The participants have a telephone visit with a study nurse after 4 and 8 week with study medication to follow-up the administration of CGRP inhibitors, headache diary and safety.

After 12 week of treatment the 3rd clinical visit is performed where the primary and secondary endpoints are registered. The participants continue to register headache diary for 4 weeks until the 3rd telephone visit which is the the end of study.

Sample size estimation: A difference of 1.6 MMDs over 12 weeks of treatment between the two groups is expected with a common standard deviation of 6.0 days for the average number of MMDs over 12 weeks in the two groups. With 90% power and a two-sided significance level of 5% 450 participants (225 in each arm) are needed in the analysis to detect the above-mentioned difference.

ELIGIBILITY:
Inclusion criteria

1. Informed and signed written consent.
2. Individuals of any sex, 18-70 years at the time of signing the informed consent.
3. Fulfilling the diagnosis chronic migraine criteria 1.3. according to the International Classification of Headache Disorders version 3 at time of inclusion.
4. Indications for treatment with CGRP mAbs according to SmPCs.
5. Indications for treatment with BTA according to SmPC.
6. No previous use of CGRP inhibitors or BTA.
7. Women of childbearing potential (WOCBP) can only be included if they use a highly effective contraception method

Exclusion criteria:

1. Contraindications, allergy or hypersensitivity reactions to BTA including infection at the injection site.
2. Contraindications, allergy or hypersensitivity reactions to CGRP mAbs including serious cardiovascular illness such as myocardial infarction, stroke, unstable angina pectoris, revascularization procedures last 12 months.
3. Concomitant medication overuse headache where drug withdrawal has not been done.
4. Subject is unable to differentiate migraine from other concomitant headaches.
5. Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months before study inclusion (Visit 2).
6. Long-standing continuous headache with no headache free days or periods for a period of time >1 years.
7. Pregnancy, planning to get pregnant, inability to use contraceptives and lactating.
8. High degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator.
9. Alcohol or illicit drug dependence.
10. Investigators may exclude patients who, for various reasons (for example, severe psychiatric disorders), are considered unlikely to be able to complete the tasks required for participation in the study.
11. Inability to understand study procedures and to comply with them for the entire length of the study, assessed at the discretion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Changer of Monthly Migraine Days over 12 weeks of treatment with the study medication. | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by reduction of Monthly Migraine Days (MMDs) over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3 - primary endpoint visit.

SECONDARY OUTCOMES:
Change of Monthly Headache Days** over 12 weeks of treatment with the study medication | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by reduction of Monthly Headache Days (MHDs) over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3.
Monthly number of days with rescue medication over 12 weeks of treatment with the study medication. | 12 weeks
  Headache diary (by using the mobile application Brain Twin) where all rescue medication is registered until Visit 3.
Number of treatment responders (≥ 50%, ≥75% and 100 % reduction in Monthly Migraine Headache days in each group over 12 weeks of treatment) at 12 weeks post-randomization. | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by number of treatment responders ≥ 50%, ≥75% and 100 % reduction in MHD and MMDs over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3.
Number of weekly migraine days from baseline to 12 months post-randomization. | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by weekly migraine days over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3.
Total number of hours at moderate or severe pain over 12 weeks of treatment. | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by total headache score per month over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3.

OTHER OUTCOMES:
Number of treatment responders (≥ 30% reduction in mean Mean Headache Days over 12 weeks of treatment) at 12 weeks post-randomization. | 12 weeks
  To assess the difference in number of treatment responders of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by difference in number of treatment responders over 12 weeks of treatment by using headache diary with the mobile application Brain Twin until assessment at Visit 3.
Number of crystal-clear headache-free days after 12 weeks of treatment with the study medication | 12 weeks.
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by number of crystal-clear headache-free days over 12 weeks of treatment using headache diary with the mobile application Brain Twin until assessment at Visit 3.
Percentage of patients fulfilling the International Classification of Headache Disorders version 3 diagnostic criteria for medication overuse headache over 12 weeks of treatment. | 12 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by change in percentage of patients fulfilling the ICHD-3 diagnostic criteria for MOH over 12 weeks of treatment. This assessment is based on information registered in the headache diary during 12 weeks and assessment at Visit 3.
Number of patients completing the trial and number of dropouts | 12 weeks.
  To assess the feasibility of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients over 12 weeks of treatment. This is assessed at Visit 3.
Change in Migraine Disability Assessment Score over 12 weeks of treatment with the study medication | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP , mAbs over 12 weeks of treatment on headache disability assessed by Migraine Disability Assessment. This questionnaire is filled in by the participant at Visit 2 and 3. Minimum Migraine Disability Assessment score 0, maximum score 270. Higher scores mean a worse outcome.
Change in Hospital Anxiety and Depression Scale score over 12 weeks of treatment with the study medication | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment on anxiety and depression. HADS-A and -D questionnaire is filled in by the participant at Visit 2 and 3. Minimum Hospital Anxiety and Depression Scale score 0, maximum value 21. Higher scores mean a worse outcome.
Change in Bergen Insomnia Scale over 12 weeks of treatment with the study medication | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment on insomnia assessed by Bergen Insomnia Scale. The questionnaire is filled in by the participant at Visit 2 and 3. Minimum Bergen Insomnia Scale Scores is 0, maximum is 42. Higher scores mean a worse outcome.
Change in Fatigue Score over 12 weeks of treatment with the study medication | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment on insomnia assessed by Bergen Insomnia Scale. The questionnaire is filled in by the participant at Visit 2 and 3. Higher scores mean a worse outcome.
Change in cognitive impairment scale for migraine attacks - Mig-SCOG score over 12 weeks of treatment with the study medication | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment on cognitive symptoms during migraine attacks assessed by subjective cognitive impairment scale for migraine attacks - Mig-SCOG score. The questionnaire is filled in by the participant at Visit 2 and 3. Minimum score 0, maximum 18. Higher scores mean a worse outcome.
Patients' Global Impression of Change scale | 12 weeks
  To assess the consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment on the patients´ global impression of change assessed by PGIC score. The questionnaire is filled in by the participant at Visit 3. Minimum Patients' Global Impression of Change scale 0, maximum 7. Higher scores mean a better outcome.
Number of days on sick leave from baseline to 12 weeks post-randomization. | 16 weeks
  To assess the efficacy of dual therapy with CGRP mAbs and BTA compared to single therapy with CGRP mAbs in chronic migraine patients measured by numbers of days of sick leave over 12 weeks of treatment. Sick leave is registered by the participant in the headache diary using the application Brain Twin and assessed at Visit 1, 2 and 3.
Costs and Quality of life measured by EuroQol 5D-5L before treatment initiation, and 12 weeks after treatment initiation | 12 weeks.
  To assess the health economic consequences of dual therapy with CGRP mAbs and BTA versus CGRP mAbs over 12 weeks of treatment. The EQ-5D-5L Questionnaire will be filled in by the participants at Visit 2 and 3.
Absenteeism from work (salary, sick leave, social security). Presenteeism (lost workplace productivity), Productivity Cost | 12 weeks
  To assess change of productivity loss over 12 weeks of treatment in the two groups by using the Institute for Medical Technology Assessment Productivity Cost Questionnaire to be filled in by the participant at Visit 3. The loading ranges from 0 to 1; the higher the value, the more an item is associated with a factor.
Assesment of resource use over 12 weeks of treatment in the two groups | 12 weeks
  Health economic assessment of resource use assessed by Norwegian Kroner.

CONTACTS AND LOCATIONS:
Locations (6):
- Norway (6):
  - Østfold Hospital Trust, Grålum
  - Sørlandet Hospital Kristiansand, Kristiansand
  - Innlandet Hospital Trust Lillehammer, Lillehammer
  - Oslo University Hospital, Oslo
  - Telemark Hospital Trust Skien, Skien
  - St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Munoz-Vendrell A, Campoy S, Caronna E, Alpuente A, Torres-Ferrus M, Nieves Castellanos C, Olivier M, Campdelacreu J, Prat J, Camina Muniz J, Molina Martinez FJ, Minguez-Olaondo A, Ruibal Salgado M, Santos Lasaosa S, Navarro Perez MP, Morollon N, Lopez Bravo A, Cano Sanchez LM, Garcia-Sanchez SM, Garcia-Ull J, Rubio-Flores L, Gonzalez-Martinez A, Quintas S, Echavarria Iniguez A, Gil Luque S, Castro-Sanchez MV, Adell Ortega V, Garcia Alhama J, Berrocal-Izquierdo N, Belvis R, Diaz-Insa S, Pozo-Rosich P, Huerta-Villanueva M. Effectiveness and safety of anti-CGRP monoclonal antibodies in patients over 65 years: a real-life multicentre analysis of 162 patients. J Headache Pain. 2023 Jun 2;24(1):63. doi: 10.1186/s10194-023-01585-2. PMID 37268904
- [Background] Zheng H, Koo EH. The amyloid precursor protein: beyond amyloid. Mol Neurodegener. 2006 Jul 3;1:5. doi: 10.1186/1750-1326-1-5. PMID 16930452
- [Background] de Vries Lentsch S, van der Arend BWH, Maassen VanDenBrink A, Terwindt GM. Blood Pressure in Patients With Migraine Treated With Monoclonal Anti-CGRP (Receptor) Antibodies: A Prospective Follow-up Study. Neurology. 2022 Oct 25;99(17):e1897-e1904. doi: 10.1212/WNL.0000000000201008. Epub 2022 Oct 4. PMID 36195452
- [Background] Chalder T, Berelowitz G, Pawlikowska T, Watts L, Wessely S, Wright D, Wallace EP. Development of a fatigue scale. J Psychosom Res. 1993;37(2):147-53. doi: 10.1016/0022-3999(93)90081-p. PMID 8463991
- [Background] Gil-Gouveia R, Oliveira AG, Martins IP. A subjective cognitive impairment scale for migraine attacks. The MIG-SCOG: development and validation. Cephalalgia. 2011 Jul;31(9):984-91. doi: 10.1177/0333102411408359. Epub 2011 May 31. PMID 21628438
- [Background] Stewart WF, Lipton RB, Whyte J, Dowson A, Kolodner K, Liberman JN, Sawyer J. An international study to assess reliability of the Migraine Disability Assessment (MIDAS) score. Neurology. 1999 Sep 22;53(5):988-94. doi: 10.1212/wnl.53.5.988. PMID 10496257
- [Background] Dodick DW, Silberstein SD, Lipton RB, DeGryse RE, Adams AM, Diener HC. Early onset of effect of onabotulinumtoxinA for chronic migraine treatment: Analysis of PREEMPT data. Cephalalgia. 2019 Jul;39(8):945-956. doi: 10.1177/0333102418825382. Epub 2019 May 21. PMID 31112399
- [Background] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019 May;39(6):687-710. doi: 10.1177/0333102419828967. Epub 2019 Feb 26. PMID 30806518
- [Background] Aurora SK, Dodick DW, Turkel CC, DeGryse RE, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT 1 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 1 trial. Cephalalgia. 2010 Jul;30(7):793-803. doi: 10.1177/0333102410364676. Epub 2010 Mar 17. PMID 20647170
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Carvalho IV, Fernandes CS, Damas DP, Barros FM, Gomes IR, Gens HM, Luzeiro I. The migraine postdrome: Clinical characterization, influence of abortive treatment and impact in the quality of life. Clin Neurol Neurosurg. 2022 Oct;221:107408. doi: 10.1016/j.clineuro.2022.107408. Epub 2022 Aug 4. PMID 35985096
- [Background] Gerstein MT, Wirth RJ, Uzumcu AA, Houts CR, McGinley JS, Buse DC, McCarrier KP, Cooke A, Touba NM, Nishida TK, Goadsby PJ, Dodick DW, Lipton RB. Patient-reported experiences with migraine-related cognitive symptoms: Results of the MiCOAS qualitative study. Headache. 2023 Mar;63(3):441-454. doi: 10.1111/head.14484. Epub 2023 Mar 10. PMID 36905166
- [Background] Lipton RB, Lanteri-Minet M, Leroux E, Manack Adams A, Contreras-De Lama J, Reed ML, Fanning KM, Buse DC. Pre- and post-headache phases of migraine: multi-country results from the CaMEO - International Study. J Headache Pain. 2023 Nov 8;24(1):151. doi: 10.1186/s10194-023-01683-1. PMID 37940856
- [Background] Khanal S, Underwood M, Naghdi S, Brown A, Duncan C, Matharu M, Mistry H. A systematic review of economic evaluations of pharmacological treatments for adults with chronic migraine. J Headache Pain. 2022 Sep 16;23(1):122. doi: 10.1186/s10194-022-01492-y. PMID 36114468
- [Background] Salim A, Hennessy E, Sonneborn C, Hogue O, Biswas S, Mays M, Suneja A, Ahmed Z, Mata IF. Synergism of Anti-CGRP Monoclonal Antibodies and OnabotulinumtoxinA in the Treatment of Chronic Migraine: A Real-World Retrospective Chart Review. CNS Drugs. 2024 Jun;38(6):481-491. doi: 10.1007/s40263-024-01086-z. Epub 2024 Apr 7. PMID 38583127
- [Background] Scuteri D, Tonin P, Nicotera P, Vulnera M, Altieri GC, Tarsitano A, Bagetta G, Corasaniti MT. Pooled Analysis of Real-World Evidence Supports Anti-CGRP mAbs and OnabotulinumtoxinA Combined Trial in Chronic Migraine. Toxins (Basel). 2022 Aug 1;14(8):529. doi: 10.3390/toxins14080529. PMID 36006191
- [Background] Ornello R, Baraldi C, Guerzoni S, Lambru G, Andreou AP, Raffaelli B, Gendolla A, Barbanti P, Aurilia C, Egeo G, Cevoli S, Favoni V, Vernieri F, Altamura C, Russo A, Silvestro M, Valle ED, Mancioli A, Ranieri A, Alfieri G, Latysheva N, Filatova E, Talbot J, Cheng S, Holle D, Scheffler A, Nezadal T, Ctrnacta D, Sipkova J, Matousova Z, Casalena A, Maddestra M, Viola S, Affaitati G, Giamberardino MA, Pistoia F, Reuter U, Sacco S. Comparing the relative and absolute effect of erenumab: is a 50% response enough? Results from the ESTEEMen study. J Headache Pain. 2022 Mar 19;23(1):38. doi: 10.1186/s10194-022-01408-w. PMID 35305579
- [Background] Sacco S, Amin FM, Ashina M, Bendtsen L, Deligianni CI, Gil-Gouveia R, Katsarava Z, MaassenVanDenBrink A, Martelletti P, Mitsikostas DD, Ornello R, Reuter U, Sanchez-Del-Rio M, Sinclair AJ, Terwindt G, Uluduz D, Versijpt J, Lampl C. European Headache Federation guideline on the use of monoclonal antibodies targeting the calcitonin gene related peptide pathway for migraine prevention - 2022 update. J Headache Pain. 2022 Jun 11;23(1):67. doi: 10.1186/s10194-022-01431-x. PMID 35690723
- [Background] Detke HC, Goadsby PJ, Wang S, Friedman DI, Selzler KJ, Aurora SK. Galcanezumab in chronic migraine: The randomized, double-blind, placebo-controlled REGAIN study. Neurology. 2018 Dec 11;91(24):e2211-e2221. doi: 10.1212/WNL.0000000000006640. Epub 2018 Nov 16. PMID 30446596
- [Background] Ferrari MD, Diener HC, Ning X, Galic M, Cohen JM, Yang R, Mueller M, Ahn AH, Schwartz YC, Grozinski-Wolff M, Janka L, Ashina M. Fremanezumab versus placebo for migraine prevention in patients with documented failure to up to four migraine preventive medication classes (FOCUS): a randomised, double-blind, placebo-controlled, phase 3b trial. Lancet. 2019 Sep 21;394(10203):1030-1040. doi: 10.1016/S0140-6736(19)31946-4. Epub 2019 Aug 16. PMID 31427046
- [Background] Tepper S, Ashina M, Reuter U, Brandes JL, Dolezil D, Silberstein S, Winner P, Leonardi D, Mikol D, Lenz R. Safety and efficacy of erenumab for preventive treatment of chronic migraine: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jun;16(6):425-434. doi: 10.1016/S1474-4422(17)30083-2. Epub 2017 Apr 28. PMID 28460892
- [Background] Silberstein SD, Dodick DW, Bigal ME, Yeung PP, Goadsby PJ, Blankenbiller T, Grozinski-Wolff M, Yang R, Ma Y, Aycardi E. Fremanezumab for the Preventive Treatment of Chronic Migraine. N Engl J Med. 2017 Nov 30;377(22):2113-2122. doi: 10.1056/NEJMoa1709038. PMID 29171818
- [Background] Corasaniti MT, Bagetta G, Nicotera P, Tarsitano A, Tonin P, Sandrini G, Lawrence GW, Scuteri D. Safety of Onabotulinumtoxin A in Chronic Migraine: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Toxins (Basel). 2023 May 12;15(5):332. doi: 10.3390/toxins15050332. PMID 37235366
- [Background] Silberstein SD, Blumenfeld AM, Cady RK, Turner IM, Lipton RB, Diener HC, Aurora SK, Sirimanne M, DeGryse RE, Turkel CC, Dodick DW. OnabotulinumtoxinA for treatment of chronic migraine: PREEMPT 24-week pooled subgroup analysis of patients who had acute headache medication overuse at baseline. J Neurol Sci. 2013 Aug 15;331(1-2):48-56. doi: 10.1016/j.jns.2013.05.003. Epub 2013 Jun 19. PMID 23790235
- [Background] Aurora SK, Dodick DW, Diener HC, DeGryse RE, Turkel CC, Lipton RB, Silberstein SD. OnabotulinumtoxinA for chronic migraine: efficacy, safety, and tolerability in patients who received all five treatment cycles in the PREEMPT clinical program. Acta Neurol Scand. 2014 Jan;129(1):61-70. doi: 10.1111/ane.12171. Epub 2013 Sep 20. PMID 24107267
- [Background] Dodick DW, Turkel CC, DeGryse RE, Aurora SK, Silberstein SD, Lipton RB, Diener HC, Brin MF; PREEMPT Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: pooled results from the double-blind, randomized, placebo-controlled phases of the PREEMPT clinical program. Headache. 2010 Jun;50(6):921-36. doi: 10.1111/j.1526-4610.2010.01678.x. Epub 2010 May 7. PMID 20487038
- [Background] Diener HC, Dodick DW, Aurora SK, Turkel CC, DeGryse RE, Lipton RB, Silberstein SD, Brin MF; PREEMPT 2 Chronic Migraine Study Group. OnabotulinumtoxinA for treatment of chronic migraine: results from the double-blind, randomized, placebo-controlled phase of the PREEMPT 2 trial. Cephalalgia. 2010 Jul;30(7):804-14. doi: 10.1177/0333102410364677. Epub 2010 Mar 17. PMID 20647171
- [Background] Blumenfeld A, Silberstein SD, Dodick DW, Aurora SK, Turkel CC, Binder WJ. Method of injection of onabotulinumtoxinA for chronic migraine: a safe, well-tolerated, and effective treatment paradigm based on the PREEMPT clinical program. Headache. 2010 Oct;50(9):1406-18. doi: 10.1111/j.1526-4610.2010.01766.x. PMID 20958294
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Steiner TJ, Stovner LJ, Vos T, Jensen R, Katsarava Z. Migraine is first cause of disability in under 50s: will health politicians now take notice? J Headache Pain. 2018 Feb 21;19(1):17. doi: 10.1186/s10194-018-0846-2. No abstract available. PMID 29468450
- [Background] GBD 2016 Headache Collaborators. Global, regional, and national burden of migraine and tension-type headache, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2018 Nov;17(11):954-976. doi: 10.1016/S1474-4422(18)30322-3. PMID 30353868
- [Background] Ashina M, Katsarava Z, Do TP, Buse DC, Pozo-Rosich P, Ozge A, Krymchantowski AV, Lebedeva ER, Ravishankar K, Yu S, Sacco S, Ashina S, Younis S, Steiner TJ, Lipton RB. Migraine: epidemiology and systems of care. Lancet. 2021 Apr 17;397(10283):1485-1495. doi: 10.1016/S0140-6736(20)32160-7. Epub 2021 Mar 25. PMID 33773613
- [Background] Mechtler L, Saikali N, McVige J, Hughes O, Traut A, Adams AM. Real-World Evidence for the Safety and Efficacy of CGRP Monoclonal Antibody Therapy Added to OnabotulinumtoxinA Treatment for Migraine Prevention in Adult Patients With Chronic Migraine. Front Neurol. 2022 Jan 6;12:788159. doi: 10.3389/fneur.2021.788159. eCollection 2021. PMID 35069416
- [Background] Pellesi L, Do TP, Ashina H, Ashina M, Burstein R. Dual Therapy With Anti-CGRP Monoclonal Antibodies and Botulinum Toxin for Migraine Prevention: Is There a Rationale? Headache. 2020 Jun;60(6):1056-1065. doi: 10.1111/head.13843. Epub 2020 May 21. PMID 32437038
- [Background] Lipton RB, Goadsby PJ, Smith J, Schaeffler BA, Biondi DM, Hirman J, Pederson S, Allan B, Cady R. Efficacy and safety of eptinezumab in patients with chronic migraine: PROMISE-2. Neurology. 2020 Mar 31;94(13):e1365-e1377. doi: 10.1212/WNL.0000000000009169. Epub 2020 Mar 24. PMID 32209650
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/